CLINICAL TRIAL: NCT06288594
Title: Assessing the Feasibility, Acceptability, and Preliminary Efficacy of the 'TraumaRelief' App for PTSD Symptom Management in Turkey: A Pilot Randomized Controlled Trial
Brief Title: TraumaRelief App: A Pilot RCT Assessing Feasibility and Acceptability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hasan arslan, Research Assistant, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEU-PSI-HA-001
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Post-Traumatic Stress Disorder (PTSD)
Keywords: Ptsd; Trauma; Mobile Application; Pilot study; Randomized Controlled Trial; Feasibility; Acceptability; Efficacy; E-health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a three-arm, parallel randomized controlled trial. Upon enrollment, participants are randomly assigned to one of three groups. The first group will use the "TraumaRelief" application in addition to weekly video calls with a psychologist. The second group will use the "TraumaRelief" mobile application exclusively. The third group will serve as a control and receive no intervention. The primary outcomes will be measured at baseline, five weeks, one month, and three months post-intervention to assess the efficacy and acceptability of the mobile application and the added benefit of psychological support.
Masking Description: In this pilot randomized controlled trial, no masking is applied, as the nature of the interventions makes it impractical. Participants are informed of their group assignment since those in the second group are aware of their additional video call sessions with psychotherapists. The therapists conducting the sessions also need to be aware of the intervention they are delivering to properly adhere to the treatment protocol. This open-label approach is necessary to facilitate the intended psychotherapeutic interactions and to ensure that the intervention is delivered with fidelity, as per the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Application Plus Online Therapist Support Group (Experimental): Participants in this arm will engage with the "TraumaRelief" mobile application while also receiving weekly online therapy sessions lasting 20 to 30 minutes for the duration of five weeks.
  Interventions: Behavioral: Application Plus Online Therapist Support Group
- Application Only Group (Experimental): Participants in this arm will utilize the "TraumaRelief" mobile application as the sole intervention over a period of five weeks. This group will not receive any therapist-led sessions or additional support outside of the application's features.
  Interventions: Behavioral: Application Only Group
- Waitlist Control Group (No Intervention): Participants in this control group are placed on a waitlist and will not receive any intervention during the initial five-week active phase of the trial. They serve as a comparative benchmark against the experimental groups to assess the effectiveness of the interventions. Following the three-month follow-up period, participants in this group will be granted access to the "TraumaRelief" mobile application, allowing them to benefit from the application.

INTERVENTIONS:
Behavioral: Application Plus Online Therapist Support Group — Participants in the therapist-supported group will receive weekly 20-30 minute online sessions for five weeks, with content based on a semi-structured manual. After 80% completion of the psychoeducation module, the coping module becomes available, and similarly, the exposure module follows. These sessions will be conducted in adherence to a structured manual, with the therapist introducing the module of the week, guiding through exercises, assigning homework, and reviewing the previous assignments. Sessions include module introductions, exercises, homework assignments, and application use review. Feedback and PCL-5 scores guide post-session recommendations. A random 40% of sessions will undergo fidelity checks by doctoral-level psychologists.
  Arms: Application Plus Online Therapist Support Group
Behavioral: Application Only Group — Participants allocated to this group will have access to the "TraumaRelief" mobile application over a five-week period, with the exception of the online module component. The application's deployment strategy ensures a structured progression through its features: participants will gain access to the subsequent modules only after completing 80% of the preceding module. Initially, they will engage with the psychoeducation module; upon completion of at least 80% of this module, the coping with symptoms module will become available. Similarly, successful engagement with 80% of the coping module will unlock the imaginary exposure module. This sequential module access is designed to reinforce the acquisition of knowledge and skills in a stepwise manner, paralleling the structure provided to the "TraumaRelief Mobile Application with Therapist Support" group, yet without the additional therapist interaction.
  Arms: Application Only Group

SUMMARY:
The world experiences a high rate of traumatic events. Even if PTSD is not diagnosed, traumatic events can significantly affect people's lives. Traditional face-to-face therapies often face challenges, such as financial constraints, expensive therapy sessions, time restrictions, fear of stigma, and difficulties in accessing clinical psychologists. These challenges motivated us to develop new methods. Particularly in Turkey, there is neither sufficient infrastructure nor existing applications dedicated to addressing trauma-related complications. The development of the 'TraumaRelief' app is a pioneering initiative aimed at bridging this gap, targeting the resolution of these prevalent issues by introducing an accessible, innovative solution. The newly developed "TraumaRelief" app aims to provide solutions to these issues. This app contains eight modules: online video talks, psychoeducation, coping with symptoms, mindfulness-based relaxation exercises, imagery exposure, CBT (Cognitive Behavioral Therapy)-based daily exercises, therapist messaging, emergency contact access. The purpose of this study is to test the feasibility and acceptability of this newly developed application through a pilot randomized controlled trial.

DETAILED DESCRIPTION:
"TraumaRelief" consists of eight modules. These are:

1. Psychoeducation Module: This module addresses fundamental questions-What is trauma? What is PTSD? What are the symptoms of PTSD?-and elaborates on related problems such as sleep, nutrition, and anger. It is designed to provide comprehensive information and guidance on these issues and comprises 10,000 words and eight animated videos (approximately 40 minutes in total).
2. Coping with Symptoms Module: This module offers 10,000 words and six animations (around 40 minutes in total) featuring information and exercises tailored to manage PTSD and related issues.
3. Imaginary Exposure Module: The module including 4,000 words and two audio recordings details the concept of imaginary exposure. The elements of this exposure are the creation of a list of avoided and uncomfortable situations, and of an hierarchy of fear, alongside instructions for imaginary exposure to avoided objects and the traumatic event itself.
4. Daily Exercises: Featuring 14 distinct audio recordings-ranging from relaxation, body scanning, breathing exercises, positive visualization, thought awareness, to compassion (each recording varies between 5 and 17 minutes)-this module integrates exercises such as automatic thought questioning and reviews, daily activity forms, and an enjoyable activity list, as directed in the coping with symptoms module.
5. Online Meeting Module: Facilitates video calls with psychologists via phone or e mail, enhancing therapeutic engagement.
6. Messaging with the Therapist: This module enables participants to send messages to their therapists through the application in emergency situations, ensuring timely support.
7. Myself Module: Each time users access the psychoeducation and coping with symptoms modules, they assess their stress level, contributing to a personalized stress graph.
8. Emergency Module: Provides contact information for relevant institutions in high-risk scenarios, such as suicidal ideation, facilitating immediate assistance.

Application Usage Pattern: Post-registration, access to subsequent modules is contingent upon the completion of prior ones, ensuring a structured progression through the content. For instance, the Imaginary Exposure Module is unlocked only after completing at least eighty percent of the Psychoeducation Module, ensuring participants have a foundational understanding before proceeding.

This pilot randomized controlled study aims to evaluate the feasibility, acceptability, and preliminary efficacy of the "TraumaRelief" application for individuals who have experienced traumatic events. The research primarily focuses on measuring application compliance and user satisfaction through metrics such as attrition, recruitment, retention, consent, adherence rates, and usage frequency. It also seeks to gather initial data on the application's impact on clinical outcomes, including PTSD symptom severity, depressive symptoms, anxiety levels, and quality of life. The procured data will provide information for designing a larger-scale RCT (Randomized Controlled Trial) and underpin subsequent efforts to refine the "TraumaRelief" application.

ELIGIBILITY:
Inclusion Criteria:

* Minimum Education Level: Participants are required to have at least a primary school education to ensure comprehension of the study materials.
* Smartphone Ownership
* Regular Smartphone Access
* PTSD Diagnosis Risk: Participants must have a PCL-5 score at or above the diagnostic threshold of 31, indicative of PTSD.

Exclusion Criteria:

* Risk of Suicide
* Neurological or Psychiatric Conditions: Participants should not have neurological or psychiatric conditions that would impede the use of the "TraumaRelief" mobile application.
* Current Medication Use: Participants who are on psychotropic medications that could influence the study's outcomes will be excluded to prevent interactions with the intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants of any gender identity are eligible to enroll in this study, reflecting our commitment to inclusivity and recognition of the diversity of gender experiences.
Enrollment: 107 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
PTSD Symptom Severity | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  This outcome measure will assess the change in severity of PTSD symptoms, utilizing the PTSD Checklist for DSM-5 (PCL-5). This self-report measure encompasses 20 items distributed across four domains: re-experiencing (comprising five items), avoidance (encompassing two items), negative alterations in cognition and mood (consisting of seven items), and hyperarousal (incorporating six items). The scoring spectrum extends from 0 to 80, with ascending scores indicative of augmented severity in PTSD symptoms. The threshold of concern has been established at 31 points. In the context of the Turkish adaptation study, the Cronbach's alpha reliability coefficient was ascertained to be .94. The instrument mandates participants to specify a particular traumatic event at the outset, thereby rendering the PCL-5 applicable for evaluating PTSD across diverse traumatic experiences.

SECONDARY OUTCOMES:
Depression Anxiety and Stress Symptom Severity | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  This measure will evaluate the change in severity of depression, anxiety, and stress symptoms, as measured by the Depression, Anxiety, and Stress Scale (DASS-21). which includes 21 items divided equally among three subscales: depression (seven items), anxiety (seven items), and stress (seven items). The scoring range is from 0 to 42 for each subscale, with higher scores denoting more significant levels of depression, anxiety, and stress. The Turkish version of the scale has demonstrated robust psychometric properties, with Cronbach's alpha internal consistency coefficients reported as .92 for the depression subscale, .86 for the anxiety subscale, and .88 for the stress subscale. This measurement tool is crucial for identifying the severity and range of these symptoms in individuals, contributing to a comprehensive understanding of their psychological well-being.
Quality of Life Improvement | Change from baseline assessment, at 1 week post-intervention assessment (6-7 weeks after baseline), change from post-assessment at 1 month post-intervention assessment (2.5-3 months after baseline), and change from at 3 month post intervention assessment
  The change in quality of life will be assessed using the [Quality of Life Scale], a validated scale for measuring various domains of life quality in individuals with PTSD. It includes 16 items, measures various domains of life quality including physical and psychological well-being, independence, social relationships, environmental factors, and spirituality among individuals with PTSD. The scoring range extends from 16 to 112, where higher scores denote an enhanced perception of life quality across these domains. The Turkish adaptation of the QOLS has demonstrated robust reliability and validity, with a Cronbach's alpha coefficient of .92, indicating a high level of internal consistency.
Feasibility: Attrition Rate | Attrition rate will be measured from baseline, at 5 weeks post-intervention, 1 month post-intervention, and 3 months post-intervention.
  The attrition rate will reflect the percentage of participants who drop out of the study at various points. This measure will help to assess the engagement and commitment levels of participants to the study protocol.
Feasibility: Recruitment Rate | Recruitment period will be calculated from the beginning of the enrollment process up to the start date of the intervention
  Recruitment rate will be calculated based on the number of participants successfully enrolled in the study over the total recruitment period. This metric will evaluate the effectiveness of the recruitment strategies used.
Feasibility: Retention Rate | Retention rate will be assessed from baseline, at 5 weeks, 1 month post-intervention, and 3 months post-intervention.
  Retention rate will be monitored to determine the proportion of participants who complete the study without dropping out. This outcome will provide insight into the sustainability and practicality of the study design.
Feasibility: Adherence Rate to the Mobile Application | Throughout the 5-week intervention period
  Adherence rate will be measured by the frequency and consistency of participants' interactions with the "TraumaRelief" mobile application. Usage data will be collected to assess how well participants stick to the prescribed intervention.
Feasibility: Consent Rate | Consent rate will be recorded from the onset of the recruitment period until the start date of the intervention.
  Consent rate will be determined by the ratio of individuals who agree to participate after being approached for the study to the total number of individuals approached, providing insight into the willingness of potential participants to engage in the study.
Feasibility: Fidelity of Intervention Delivery | Throughout the 5-week intervention period
  To assess the fidelity of the delivered intervention, 40% of the therapy sessions conducted via video calls will be randomly selected and evaluated by clinical psychologists who have completed their doctoral studies in the field. These sessions will be scored using a fidelity checklist to ensure that the intervention is being administered as per the established protocol. This process will help maintain the quality and consistency of the intervention across all participants.
Acceptability: System Usability Scale (SUS) Score for Acceptability | End of the 5-week intervention period
  The acceptability of the "TraumaRelief" mobile application among participants will be measured using the System Usability Scale (SUS) score. This 10-item questionnaire is a well-established method for assessing system usability, employing a scoring range from 0 to 100. Higher SUS scores are indicative of enhanced usability, suggesting a more user-friendly interface and satisfactory user interaction, thus reflecting the application's overall acceptability. The SUS-TR, tailored for the Turkish context , demonstrated high reliability among a sample of 324 university students. The scoring methodology allows for scores to be interpreted along a continuum, where higher values denote greater system usability and user satisfaction, affirming the scale's validity and reliability for Turkish users.
Acceptability: Preferred and Least Preferred Module Components | End of each module during the 5-week intervention period
  Participants will report the components they found most and least beneficial within each module. This feedback will be used to gauge the acceptability and to refine module content to enhance user experience and engagement
Acceptability: Application Utilization Frequency | Daily throughout the 5-week intervention period
  Usage frequency will be assessed by the average daily number of times participants engage with the "TraumaRelief" application. This metric reflects the integration of the app into daily routines, indicating its acceptability and practicality.
Acceptability: Likelihood to Recommend the Application | At the end of the 5-week intervention period
  The likelihood of participants recommending the "TraumaRelief" application to someone they care about will be measured. A high likelihood of recommendation will indicate the intervention's acceptability and potential endorsement by users.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan ARSLAN, PHD. Cand., Principal Investigator — Dokuz Eylul University; A. Esin YILMAZ SAMANCI, professor, Study Director — Dokuz Eylul University
Locations (1):
- Hasan arslan, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arslan H, Yilmaz AE. Assessing the feasibility, acceptability, and preliminary efficacy of the 'TraumaRelief' app for PTSD symptom management in Turkey: Study protocol for a pilot randomized controlled trial. Internet Interv. 2024 Nov 23;38:100793. doi: 10.1016/j.invent.2024.100793. eCollection 2024 Dec. PMID 39659870